CLINICAL TRIAL: NCT05982743
Title: A Pilot Study of Using Fermented Milk Containing Lactobacillus Casei Strain Shirota (LcS) in Some Constipated Adults Having High Prevalence of Hard Stools in Vietnam
Brief Title: Lactobacillus Casei Strain Shirota Fermented Milk for Alleviating Hard Stools in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult Honsha Co., LTD (Industry)
Collaborators: Bach Mai Hospital (Other); Vietnam National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAK-VN-001
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented milk drink (Experimental)
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota fermented milk
- No drink (No Intervention)

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei strain Shirota fermented milk — Participants will take one bottle (65 ml) of Yakult® drink daily, containing at least 6.5 x 10^9 CFU of Lactobacillus casei strain Shirota, for a period of 4 weeks. Subsequently, there will be a two-week follow-up period.
  Arms: Fermented milk drink

SUMMARY:
The objective of this study is to provide evidence supporting the efficacy of fermented milk containing Lactobacillus casei strain Shirota in alleviating hard or lumpy stools. A randomized, controlled trial has been designed on constipated adults with a high prevalence of hard stools in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, aged between 18 to 60 years.
* Aware of producing hard or lumpy stools (BS score of 1 or 2) frequently.
* Produce hard or lumpy stools (BS score of 1 or 2) ≥ 25% of bowel movements during 2 weeks of screening period.
* Voluntarily provide written informed consent to participate in the study.

Exclusion Criteria:

* Subjects whose constipation symptoms are caused by primary organic disease of the colon or pelvic floora or which, in the Investigator's opinion, is caused by medication (e.g. morphine, codeine).
* Subjects with metabolic disorders, neurological disorders or any significant diseases or concomitant condition (e.g. abdominal/gastrointestinal surgery) that, in the investigator's opinion, would interfere with participation in the study.
* Subjects with any known allergic reactions to any ingredients of milk.
* Pregnant or nursing (breast-feeding) women.
* Subjects who are unable to refrain from or anticipate the use of any medication (including laxatives, diuretics, prescription and non-prescription drugs, vitamins and herbal supplements), except for paracetamol, oral contraceptives, or hormonal replacement therapy from 2-week before the initiation of screening of subject BS score to the end of the study.
* Subjects who are unable to refrain from or anticipate the use of any probiotics, prebiotics or yogurts from 2-week before the initiation of screening of subject BS score to the end of the study.
* Participation in another study with Investigational product within 2 months prior to this study.
* Drug or alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that produce hard or lumpy stools (Bristol stool form scale (BS) score of 1 or 2) ≥ 25% of bowel movements | During four weeks from the date of the site visit to submit a baseline stool sample.
  Overall treatment effect during the intervention period will be estimated using mixed effects logistic regression (with a random intercept) which include "Groups (Yakult/non-treatment)", "Weeks (first/second two weeks of the intervention period)", "baseline (median BS score during baseline)" and "Gender (women/men)" as the independent variables. "Groups x Weeks" interaction will not be included because it was absent in the past RCT studies giving Yakult.

SECONDARY OUTCOMES:
Stool frequency with hard or lumpy one (BS score of 1 or 2) | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency with ideal stool (BS score of 4) | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency, as measured by a daily stool diary | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency with straining during evacuation, as measured by a daily stool diary (Yes/No) | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency with sensation of remaining stool in the rectum after the evacuation, as measured by a daily stool diary (Yes/No) | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency with sensation of anorectal blockage, as measured by a daily stool diary (Yes/No) | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool frequency with which manual maneuvers are used, as measured by a daily stool diary (Yes/No) | During four weeks from the date of the site visit to submit a baseline stool sample.
Chinese Constipation Questionnaire score | During four weeks from the date of the site visit to submit a baseline stool sample.
Stool microbiota (increase in the abundance of bifidobacteria) | During four weeks from the date of the site visit to submit a baseline stool sample.

OTHER OUTCOMES:
BS score of the first stool after waking up (descriptive analysis) | During four weeks from the date of the site visit to submit a baseline stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: Vinh Van Hoang, PhD, Principal Investigator — Vietnam National University
Locations (1):
- Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No